CLINICAL TRIAL: NCT03393013
Title: A Phase 1b/2 Study of KZR-616 in Patients With Systemic Lupus Erythematosus With and Without Nephritis (MISSION)
Brief Title: A Study of KZR-616 in Patients With SLE With and Without Lupus Nephritis
Acronym: MISSION
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kezar Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KZR-616-002
Record Dates: First submitted 2017-12-21; First posted 2018-01-08 (Actual); Results first posted 2024-03-08 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Lupus Nephritis; Systemic Lupus Erythematosus
Keywords: immunoproteasome inhibition; selective proteasome inhibition; proteasome; lupus nephritis; lupus; nephritis; active proliferative lupus nephritis; open-label; systemic lupus erythematosus; lupus erythematosus
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic; Nephritis | interventions — KZR-616

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- KZR-616 45 mg + standard of care therapy (Phase 1b) (Experimental): Dose escalation cohort of patients with SLE with and without nephritis to receive 45 mg dose level of KZR-616 in combination with standard of care therapy.
  Two Phase 1b cohorts received 45 mg at some point during the study.
  Cohort 1 received 45 mg zetomipzomib frozen maleate weekly for 13 weeks.
  Cohort 2a followed a step-up dosing procedure. Patients received zetomipzomib frozen maleate, 30 mg weekly for 2 weeks, followed by 45 mg weekly for 2 weeks then followed by 60 mg weekly for 9 weeks.
  KZR-616 was administered as a SC injection.
  Interventions: Drug: KZR-616
- KZR-616 60 mg + standard of care therapy (Phase 1b) (Experimental): Dose escalation cohort of patients with SLE with and without nephritis to receive 60 mg dose level of KZR-616 in combination with standard of care therapy.
  Four Phase 1b cohorts received 60 mg at some point during the study.
  Cohort 2 received 60 mg zetomipzomib frozen maleate weekly for 13 weeks.
  Cohorts 2a, 2b, and 2c all followed a step-up dosing procedure. Patients in Cohort 2a received zetomipzomib frozen maleate, 30 mg weekly for 2 weeks, followed by 45 mg weekly for 2 weeks then followed by 60 mg weekly for 9 weeks. Patients in Cohort 2b received zetomipzomib lyophile, 30 mg weekly for 1 week, followed by 60 mg weekly for 12 weeks. Patients in Cohort 2c (tolerability strategies cohort) received zetomipzomib lyophile, 30 mg weekly for 1 week, followed by 60 mg weekly for 12 weeks.
  KZR-616 was administered as a SC injection.
  Interventions: Drug: KZR-616
- KZR-616 75 mg + standard of care therapy (Phase 1b) (Experimental): Dose escalation cohort of patients with SLE with and without nephritis to receive 75 mg dose level of KZR-616 in combination with standard of care therapy.
  One Phase 1b cohort received 75 mg at some point during the study.
  Cohort 3 followed a step-up dosing procedure. Patients in Cohort 3 received zetomipzomib lyophile, 30 mg weekly for 1 week, followed by 75 mg weekly for 12 weeks.
  KZR-616 was administered as a SC injection.
  Interventions: Drug: KZR-616
- KZR-616 60 mg + standard therapy (Phase 2) (Experimental): 60 mg dose level of KZR-616 selected based on data from the phase 1b dose escalation and administered to patients with active lupus nephritis in combination with standard therapy including at least one immunosuppressive agent.
  KZR-616 was administered as a SC injection weekly at a dose of 60 mg for 24 weeks (including a step-up from an initial Week 1 dose of 30 mg).
  ** See Limitations/Caveats for additional information
  Interventions: Drug: KZR-616

INTERVENTIONS:
Drug: KZR-616 — Subcutaneous Injection of KZR-616
  Other Names: zetomipzomib

SUMMARY:
This was a Phase 1b/2, multi-center study in which patients received KZR-616, administered as a subcutaneous (SC) injection weekly for 13 weeks (Phase 1b) or 24 weeks (Phase 2).

DETAILED DESCRIPTION:
This was a Phase 1b/2, open-label, multi-center study in which patients received zetomipzomib administered as a SC injection weekly for either 13 weeks (Phase 1b) or for 24 weeks (Phase 2). In both phases, safety assessments continued for up to 12 weeks following the last dose of zetomipzomib.

Phase 1b was an open-label, multiple dose escalation study designed to evaluate the safety and tolerability of escalating doses of zetomipzomib when administered in addition to standard-of-care therapy in patients with SLE with or without nephritis. For each cohort, at least 6 patients were to be enrolled to assure the availability of at least 4 evaluable patients. Decisions to escalate, expand, or decrease the dose level or dosing frequency following the first 4 weeks of dosing for at least 4 evaluable patients in a cohort were made following review by a data monitoring committee (DMC).

The zetomipzomib formulations and doses administered by cohort in Phase 1b were:

* Cohort 1: zetomipzomib frozen maleate, 45 mg weekly × 13 weeks
* Cohort 2: zetomipzomib frozen maleate, 60 mg weekly × 13 weeks
* Cohort 2a: zetomipzomib frozen maleate, 30 mg weekly × 2 weeks, followed by 45 mg weekly × 2 weeks, followed by 60 mg weekly × 9 weeks
* Cohort 2b: zetomipzomib lyophile, 30 mg weekly × 1 week, followed by 60 mg weekly × 12 weeks
* Cohort 2c: zetomipzomib lyophile, 30 mg weekly × 1 week, followed by 60 mg weekly × 12 weeks (tolerability strategies cohort)
* Cohort 3: zetomipzomib lyophile, 30 mg weekly × 1 week, followed by 75 mg weekly × 12 weeks

The Phase 2 portion of the open-label study was designed to evaluate the renal response, safety, and tolerability of a single dose level (60 mg) of zetomipzomib administered weekly in addition to standard therapy in patients with active proliferative lupus nephritis (LN) (Class III or IV, with or without Class V disease) with a UPCR ≥1.0. Patients must have been on standard therapy for LN including at least 1 immunosuppressive agent. Zetomipzomib was administered as a SC injection weekly for 24 weeks (including a step up from an initial Week 1 dose of 30 mg).

ELIGIBILITY:
Key Inclusion Criteria:

Phase 1b:

* Fulfilled the 2012 Systemic Lupus International Collaborating Clinics (SLICC) classification for SLE
* Had a positive antinuclear antibody (ANA) titer, anti-double stranded DNA (dsDNA) antibody titer, or a positive anti-Smith antibody titer
* Had active SLE (as indicated by Systemic Lupus Erythematosus Disease Activity Index 2000 [SLEDAI-2K] score ≥4), and
* Had received at least 1 prior therapy for SLE

Phase 2:

* Had active proliferative LN (Class III or IV, with or without Class V disease)
* Had a UPCR ≥1.0 measured in 24-hour urine collection
* Had a histologic diagnosis of LN on renal biopsy within the prior 2 years; for biopsies > 1 year before the Screening visit, one of the following must also be present at screening: low C3, low C4, or anti-ds-DNA elevated to above normal range
* Fulfilled the 2012 SLICC classification for SLE
* Had a positive ANA titer, anti-dsDNA antibody titer, or anti-Smith antibody titer, and
* Were currently receiving ≥1 immunosuppressive agent at a stable dose and route of administration for ≥8 weeks. If the patient is also on corticosteroids then must be on a stable dose for ≥ 2 weeks prior to Baseline

Key Exclusion Criteria:

Phase 1b:

* Current or medical history of:

  * Central nervous system manifestations by autoimmune disease
  * Overlapping autoimmune condition that may affect study assessments/outcomes
  * Antiphospholipid syndrome with history of thromboembolic event of within the 52 weeks prior to Screening
  * Malignancy of any type, with exceptions for in situ cancer that has been completely excised and certain cancers >5 years ago
* Positive test at Screening for HIV, hepatitis B/C
* Major surgery within 4 weeks before signing informed consent form or planned major surgery during the study period

Phase 2:

* Current or medical history of:

  * Central nervous system manifestations of SLE
  * Overlapping autoimmune condition that may affect study assessments/outcomes
  * Antiphospholipid syndrome with history of thromboembolic event of within the 52 weeks prior to Screening
  * Malignancy of any type within the last 5 years, with exceptions for appropriately excised and cured cervical carcinoma in situ or excised basal or squamous cell carcinomas of the skin
* Has received dialysis within the 52 weeks prior to Screening
* Positive test at Screening for HIV, hepatitis B/C
* Major surgery within 12 weeks before signing informed consent form or planned major surgery during the study period
* Use of investigational therapy or device, and/or participation in an investigational trial <8 weeks or 5 half-lives, whichever is longer, prior to Baseline; Patients who participated in Phase 1b of KZR-616-002 are excluded from Phase 2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kezar, Study Director — Kezar Life Sciences, Inc.
Locations (36):
- United States (17):
  - Academic Medical Research Institute, Los Angeles, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - SouthCoast Research Center, Inc., Miami, Florida
  - Hope Clinical Trials, Inc., Miami, Florida
  - Omega Research Maitland, Orlando, Florida
  - Arthritis Center, Inc, Palm Harbor, Florida
  - Advent Health Medical Group, Tampa, Florida
  - University of Iowa, Iowa City, Iowa
  - Northwell Health, Great Neck, New York
  - NYU Langone Orthopedic Center - Seligman Center for Advanced Therapeutics, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - SC Nephrology & Hypertension Center, Inc., Orangeburg, South Carolina
  - Ramesh C. Gupta, MD, Memphis, Tennessee
  - MedResearch, Inc., El Paso, Texas
  - Accurate Clinical Research, Inc., Houston, Texas
  - Accurate Clinical Management, LLC, Houston, Texas
- Australia (2):
  - Monash Health, Clayton, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Colombia (5):
  - Centro Integral de Reumatologia de Caribe CIRCARIBE S.A.S, Barranquilla, Atlántico
  - Clinica de la Costa, Barranquilla, Atlántico
  - Medicity SAS, Santander, Bucaramanga
  - Servimed S.A.S., Bucaramanga, Santander Department
  - Clinica de Artritis Temprana, Cali, Valle del Cauca Department
- Mexico (4):
  - Centro Integral de Reumatologia SA de CV, Guadalajara, Jalisco
  - Hospital Universitario Dr José Eleuterio Gonzalez, Monterrey, Nuevo León
  - Instituto Nacional de Cardiología Ignacio Chavez, Mexico City
  - Instituto Nacional de Ciencias Médicas y Nutricion "Salvador Zubiran", Mexico City
- Peru (3):
  - Centro de Investigación Clínica Trujillo E.I.R.L/ Clínica Peruano Americana S.A., Trujillo, La Libertad
  - Investigaciones Clinicas SAC, Lima
  - Unidad de Investigacion en Reumatologia e Inmunologia Clinica San Juan Bautista, Lima
- Bioclinica, Lodz, Poland
- Russia (3):
  - Kuzbass Clinical Hospital, Kemerovo
  - Medical Center Revma-Med, Kemerovo
  - Tolyatti City Clinical Hospital #1, Tolyatti
- Harmoniya Krasy, Kyiv, Kyiv Governorate, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Avasare R, Drexler Y, Caster DJ, Mitrofanova A, Jefferson JA. Management of Lupus Nephritis: New Treatments and Updated Guidelines. Kidney360. 2023 Oct 1;4(10):1503-1511. doi: 10.34067/KID.0000000000000230. PMID 37528520
- See also: Kezar Life Sciences, Inc. corporate website — https://www.kezarlifesciences.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who were enrolled in Phase 1b were ineligible to enroll in the Phase 2 portion of the study.
Groups:
- Cohort 1, KZR-616 QW, 45 mg + SOC (Phase 1b): Dose escalation cohort of patients with SLE with and without nephritis to receive KZR-616 45 mg once weekly (QW) for 13 weeks in combination with standard of care (SOC) therapy.
  KZR-616: Subcutaneous Injection of KZR-616
- Cohort 2, KZR-616 QW, 60 mg + SOC (Phase 1b): Dose escalation cohort of patients with SLE with and without nephritis to receive KZR-616 60 mg QW for 13 weeks in combination with SOC therapy.
  KZR-616: Subcutaneous Injection of KZR-616
- Cohort 2a, KZR-616 QW, 30 mg x 2 Wks, 45 mg x 2 Wks, 60 mg x 9 Wks + SOC (Phase 1b): Dose escalation cohort of patients with SLE with and without nephritis to receive KZR-616 30 mg QW for 2 weeks, 45 mg QW for 2 weeks, and then 60 mg QW for 9 weeks in combination with SOC therapy.
  KZR-616: Subcutaneous Injection of KZR-616
- Cohort 2b, KZR-616 QW, 30 mg x 1 wk, 60 mg x 12 Wks + SOC (Phase 1b): Dose escalation cohort of patients with SLE with and without nephritis to receive KZR-616 60 mg QW (following an initial Week 1 dose of 30 mg) for 12 weeks in combination with SOC therapy.
  KZR-616: Subcutaneous Injection of KZR-616
- Cohort 2c, KZR-616 QW, 30 mg x 1 wk, 60 mg x 12 Wks + SOC (Phase 1b): Dose escalation cohort of patients with SLE with and without nephritis to receive KZR-616 60 mg QW (following an initial Week 1 dose of 30 mg) for 12 weeks in combination with SOC therapy.
  This cohort was the tolerability strategy cohort, which introduced prophylactic measures of hydration with an oral electrolyte and non-sedating antihistamines for the first two doses.
  KZR-616: Subcutaneous Injection of KZR-616
- Cohort 3, KZR-616 QW, 30 mg x 1 wk, 75 mg x 12 Wks + SOC (Phase 1b): Dose escalation cohort of patients with SLE with and without nephritis to receive KZR-616 75 mg QW (following an initial Week 1 dose of 30 mg) for 12 weeks in combination with SOC therapy.
  KZR-616: Subcutaneous Injection of KZR-616
- KZR-616 QW, 60 mg + SOC (Phase 2): KZR-616 was administered as a subcutaneous injection QW for 24 weeks (including an initial Week 1 dose of 30 mg).
  60 mg dose level of KZR-616 selected based on data from the Phase 1b dose escalation and administered to patients with active lupus nephritis in combination with SOC therapy including at least one immunosuppressive agent.
  KZR-616: Subcutaneous Injection of KZR-616
  *See Limitations/Caveats for additional information
Period: Phase 1b
Arm/Group | Cohort 1, KZR-616 QW, 45 mg + SOC (Phase 1b) | Cohort 2, KZR-616 QW, 60 mg + SOC (Phase 1b) | Cohort 2a, KZR-616 QW, 30 mg x 2 Wks, 45 mg x 2 Wks, 60 mg x 9 Wks + SOC (Phase 1b) | Cohort 2b, KZR-616 QW, 30 mg x 1 wk, 60 mg x 12 Wks + SOC (Phase 1b) | Cohort 2c, KZR-616 QW, 30 mg x 1 wk, 60 mg x 12 Wks + SOC (Phase 1b) | Cohort 3, KZR-616 QW, 30 mg x 1 wk, 75 mg x 12 Wks + SOC (Phase 1b) | KZR-616 QW, 60 mg + SOC (Phase 2)
Started | 8 | 5 | 14 | 6 | 8 | 6 | 0
Completed | 5 | 2 | 10 | 6 | 8 | 4 | 0
Not Completed | 3 | 3 | 4 | 0 | 0 | 2 | 0
Period: Phase 2
Arm/Group | Cohort 1, KZR-616 QW, 45 mg + SOC (Phase 1b) | Cohort 2, KZR-616 QW, 60 mg + SOC (Phase 1b) | Cohort 2a, KZR-616 QW, 30 mg x 2 Wks, 45 mg x 2 Wks, 60 mg x 9 Wks + SOC (Phase 1b) | Cohort 2b, KZR-616 QW, 30 mg x 1 wk, 60 mg x 12 Wks + SOC (Phase 1b) | Cohort 2c, KZR-616 QW, 30 mg x 1 wk, 60 mg x 12 Wks + SOC (Phase 1b) | Cohort 3, KZR-616 QW, 30 mg x 1 wk, 75 mg x 12 Wks + SOC (Phase 1b) | KZR-616 QW, 60 mg + SOC (Phase 2)
Started (Patients who were in Cohorts 1, 2, 2a, 2b, 2c, and 3 were enrolled in Phase 1b only.) | 0 | 0 | 0 | 0 | 0 | 0 | 22
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 18
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1, KZR-616 QW, 45 mg + SOC (Phase 1b) | Cohort 2, KZR-616 QW, 60 mg + SOC (Phase 1b) | Cohort 2a, KZR-616 QW, 30 mg x 2 Wks, 45 mg x 2 Wks, 60 mg x 9 Wks + SOC (Phase 1b) | Cohort 2b, KZR-616 QW, 30 mg x 1 wk, 60 mg x 12 Wks + SOC (Phase 1b) | Cohort 2c, KZR-616 QW, 30 mg x 1 wk, 60 mg x 12 Wks + SOC (Phase 1b) | Cohort 3, KZR-616 QW, 30 mg x 1 wk, 75 mg x 12 Wks + SOC (Phase 1b) | KZR-616 QW, 60 mg + SOC (Phase 2) | Total
Number analyzed (Participants) | 8 | 5 | 14 | 6 | 8 | 6 | 22 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (11.5) | 46.2 (11.3) | 53.6 (15.3) | 54.3 (14.8) | 48.1 (10.3) | 45.0 (17.5) | 34.6 (11.7) | 45.5 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 12 | 6 | 8 | 6 | 20 | 65
  Male | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 10 | 2 | 5 | 3 | 12 | 39
  Not Hispanic or Latino | 4 | 2 | 4 | 4 | 3 | 3 | 10 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 2 | 1 | 3 | 1 | 11
  White | 7 | 3 | 12 | 4 | 7 | 3 | 7 | 43
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 9
UPCR at Baseline [Mean (Standard Deviation); unit: mg/mg] — UPCR = urine protein to creatinine ratio
  For Phase 1b only, UPCR was measured in g/g. Population: This baseline metric was measured for all patients in Phase 2. For Phase 1b, only two patients had active lupus nephritis with significant proteinuria.
  mg/mg
    number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0 | 22 | 24
    (all) |  |  | 3.85 |  | 2.39 |  | 2.50 (2.56) | 2.55 (2.46)
eGFR Level at Baseline [Mean (Standard Deviation); unit: mL/min/1.73 m^2] — eGFR = estimated glomerular filtration rate Population: This baseline metric was only measured for patients in Phase 2. Additionally, this baseline metric is not available for one patient from Phase 2 who was enrolled in an earlier protocol amendment.
  ** See Limitations/Caveat Section
  mL/min/1.73 m^2
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 21
    (all) |  |  |  |  |  |  | 104.71 (32.579) | 104.71 (32.579)

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Patients Who Experienced at Least One Treatment-Related Treatment-Emergent Adverse Event
Description: The safety and tolerability of zetomipzomib (KZR-616) when administered as a subcutaneous injection weekly for 13 weeks in adult patients with systemic lupus erythematous (SLE) with and without nephritis, as assessed by number of patients who experienced at least one treatment-related treatment-emergent adverse event.
  For additional information about the safety and tolerability of KZR-616, please reference the adverse events section of this posting.
Time Frame: 25 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, KZR-616 QW, 45 mg + SOC (Phase 1b) | Cohort 2, KZR-616 QW, 60 mg + SOC (Phase 1b) | Cohort 2a, KZR-616 QW, 30 mg x 2 Wks, 45 mg x 2 Wks, 60 mg x 9 Wks + SOC (Phase 1b) | Cohort 2b, KZR-616 QW, 30 mg x 1 wk, 60 mg x 12 Wks + SOC (Phase 1b) | Cohort 2c, KZR-616 QW, 30 mg x 1 wk, 60 mg x 12 Wks + SOC (Phase 1b) | Cohort 3, KZR-616 QW, 30 mg x 1 wk, 75 mg x 12 Wks + SOC (Phase 1b)
Number analyzed (Participants) | 8 | 5 | 14 | 6 | 8 | 6
Participants | 7 | 5 | 11 | 3 | 6 | 3

2. Primary Outcome: Phase 2: Number of Patients With Lupus Nephritis With a 50% Reduction in UPCR
Description: To assess the number of patients with lupus nephritis with a 50% reduction in UPCR after 24 weeks of weekly SC injections with KZR-616 when compared to baseline.
Time Frame: 24 weeks
Population: Outcome only measured for Phase 2.
  One patient is excluded (N=21) due to enrollment under an earlier Protocol Amendment.
  Prior to the open-label design, 1 patient was enrolled in Phase 2. Efficacy data for this patient are not included in this analysis because the patient received zetomipzomib for a shorter time duration (13 weeks) than specified by the outcome measure.
  *See Limitations and Caveats section for more information
Measure: Count of Participants; unit: Participants
Arm/Group | KZR-616 QW, 60 mg + SOC (Phase 2)
Number analyzed (Participants) | 21
Participants | 11

3. Secondary Outcome: Phase 1b: PK of KZR-616 (Cmax)
Description: This is the maximum observed plasma concentration (Cmax) observed after administration of KZR-616 at Week 5. The PK parameters were calculated using all timepoints at which the concentration was measured, ie. predose and 5, 15, 30 minutes, 1, 2, 4, and 8 hours postdose.
Time Frame: 8 hours
Population: This outcome was only measured in Phase 1b. The PK population is different than the overall studied population. As is pre-specified in the study protocol, analysis was completed per dose/treatment instead of per cohort for PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- KZR-616 30 mg + Standard of Care Therapy: Although there was no 30 mg dose group planned for phase 1b, an arm was included for those patients that only received 30 mg as a step up dose.
  Four Phase 1b cohorts (Cohorts 2a, 2b, 2c, and 3) received 30 mg of KZR-616 at some point during the study.
  Dose level groups are determined based on last dose received.
- KZR-616 45 mg + Standard of Care Therapy (Phase 1b): Dose escalation cohort of patients with SLE with and without nephritis to receive 45 mg dose level of KZR-616 in combination with standard of care therapy.
  Two Phase 1b cohorts (Cohorts 1 and 2a) received 45 mg of KZR-616 at some point during the study.
  Dose level groups are determined based on last dose received.
  KZR-616: Subcutaneous Injection of KZR-616
- KZR-616 60 mg + Standard of Care Therapy (Phase 1b): Dose escalation cohort of patients with SLE with and without nephritis to receive 60 mg dose level of KZR-616 in combination with standard of care therapy.
  Four Phase 1b cohorts (Cohorts 2, 2a, 2b, and 2c) received 60 mg of KZR-616 at some point during the study.
  Dose level groups are determined based on last dose received.
  KZR-616: Subcutaneous Injection of KZR-616
- KZR-616 75 mg + Standard of Care Therapy (Phase 1b): Dose escalation cohort of patients with SLE with and without nephritis to receive 75 mg dose level of KZR-616 in combination with standard of care therapy.
  One Phase 1b cohort (Cohort 3) received 75 mg of KZR-616 at some point during the study.
  Dose level groups are determined based on last dose received.
  KZR-616: Subcutaneous Injection of KZR-616
Arm/Group | KZR-616 30 mg + Standard of Care Therapy | KZR-616 45 mg + Standard of Care Therapy (Phase 1b) | KZR-616 60 mg + Standard of Care Therapy (Phase 1b) | KZR-616 75 mg + Standard of Care Therapy (Phase 1b)
Number analyzed (Participants) | 1 | 9 | 20 | 4
ng/mL | 74.2 | 134 (45.6) | 151 (50.3) | 265 (60.4)

4. Secondary Outcome: Phase 1b: PK of KZR-616 (Tmax)
Description: This is the time to maximum observed plasma concentration (tmax) observed after administration of KZR-616 at Week 5. The PK parameters were calculated using all timepoints at which the concentration was measured, ie. predose and 5, 15, 30 minutes, 1, 2, 4, and 8 hours postdose.
Time Frame: 8 hours
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | KZR-616 30 mg + Standard of Care Therapy | KZR-616 45 mg + Standard of Care Therapy (Phase 1b) | KZR-616 60 mg + Standard of Care Therapy (Phase 1b) | KZR-616 75 mg + Standard of Care Therapy (Phase 1b)
Number analyzed (Participants) | 1 | 9 | 20 | 4
hours | 1.00 | 0.25 [0.13 to 1.00] | 0.25 [0.08 to 2.00] | 0.50 [0.25 to 0.52]

5. Secondary Outcome: Phase 1b: PK of KZR-616 (AUC)
Description: This is the area under the curve (AUC) from predose through 8 hour postdose observed after administration of KZR-616 at Week 5. The PK parameters were calculated using all timepoints at which the concentration was measured, ie. predose and 5, 15, 30 minutes, 1, 2, 4, and 8 hours postdose.
Time Frame: 8 hours
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/ml
Arm/Group | KZR-616 30 mg + Standard of Care Therapy | KZR-616 45 mg + Standard of Care Therapy (Phase 1b) | KZR-616 60 mg + Standard of Care Therapy (Phase 1b) | KZR-616 75 mg + Standard of Care Therapy (Phase 1b)
Number analyzed (Participants) | 1 | 8 | 19 | 4
ng*h/ml | 258 | 387 (38.1) | 430 (36.8) | 636 (31.7)

6. Secondary Outcome: Phase 2: Number of Patients With a Partial Renal Response
Description: Number of patients with a partial renal response (PRR) after 24 weeks of treatment, as defined by:
  1. For this outcome measure, Primary UPCR criterion was used (a 50% reduction of UPCR and reduction of UPCR to <1.0 if baseline UPCR was <3.0 (or reduction of UPCR to <3.0 if baseline was ≥3.0))
  2. eGFR of greater than or equal to 60 mL/min/1.73 m^2 or no worsening of eGFR from baseline of greater than or equal to 25%
  3. No use of prohibited medication
  Count of patients below includes those who satisfy all three of the above criteria.
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | KZR-616 QW, 60 mg + SOC (Phase 2)
Number analyzed (Participants) | 21
Participants | 10

7. Secondary Outcome: Phase 2: Safety and Tolerability of KZR-616 When Administered as a SC Injection Weekly for 24 Weeks
Description: Exposure adjusted adverse event incidence rate for Injection Site Reactions and Systemic Injection Reactions.
  For additional information about the safety and tolerability of KZR-616, please reference the adverse events section of this posting.
Time Frame: 37 weeks
Population: This outcome measure was only analyzed for Phase 2.
Measure: Number; unit: events per person-weeks
Units Other Than Participants: Number of exposures
Arm/Group | KZR-616 QW, 60 mg + SOC (Phase 2)
Number analyzed (Participants) | 22
Number analyzed (Number of exposures) | 447
events per person-weeks
  Injection Site Reactions | 0.036
  Systemic Injection Reactions | 0.045

8. Secondary Outcome: Phase 1b: Recommended Phase 2 Doses of Zetomipzomib When Administered as a Subcutaneous Injection
Description: The safety data from Phase 1b were used to determine a recommended dose of zetomipzomib to administer to patients with active proliferative lupus nephritis in Phase 2 of this study. As pre-specified in the study protocol, this outcome measure was to be determined qualitatively through discussion of relevant information from the Phase 1b portion of the trial at a data monitoring committee meeting.
Time Frame: 25 weeks
Population: The DMC reviewed cumulative Phase 1b study data and provided a recommendation for the Phase 2 dose.
Measure: Number; unit: mg
Groups:
- All Phase 1b Patients (Cohort 1, Cohort 2a-c, Cohort 3): The DMC reviewed the data of the Phase 1b patient population. These patients received varying doses (30, 45, 60, or 75 mg) of KZR-616 depending on their study cohort and whether their cohort had a step-up dosing procedure included.
  KZR-616: Subcutaneous Injection of KZR-616
Arm/Group | All Phase 1b Patients (Cohort 1, Cohort 2a-c, Cohort 3)
Number analyzed (Participants) | 47
mg | 60

9. Post Hoc Outcome: Phase 1b: Changes in UPCR in Patients With SLE Who Had Active Lupus Nephritis
Description: Changes in lupus disease assessments and changes from baseline in laboratory measures
  - Renal parameters (UPCR) in Patients with SLE who had active lupus nephritis at baseline, 13 weeks (end of treatment), and 25 weeks (end of study)
Time Frame: Week 25
Population: Only two patients in the Phase 1b study had active lupus nephritis.
Measure: Number; unit: g/g
Groups:
- Patient 1: Enrolled in Cohort 2a where participants received 13 weeks of KZR-616:
  - 2 weeks of 30 mg, followed by 2 weeks of 45 mg, and 9 weeks of 60 mg
- Patient 2: Enrolled in Cohort 2c where participants received 13 weeks of KZR-616:
  - 1 week of 30 mg and then 12 weeks of 60 mg
Arm/Group | Patient 1 | Patient 2
Number analyzed (Participants) | 1 | 1
g/g
  Baseline | 3.85 | 2.39
  Week 13 (End of Treatment) | 2.89 | 0.69
  Week 25 (End of Study) | 1.12 | 1.47

ADVERSE EVENTS:
Time Frame: The adverse event data was collected starting at the time of signed informed consent and were collected until 12 weeks after last dose. This time period was approximately 25 and 37 weeks for each participant in Phase 1b and Phase 2, respectively.
Description: Anticipated fluctuations of pre-existing conditions, including the disease under study, that do not represent a clinically significant exacerbation or worsening need not be considered AEs.
Arm/Group | Cohort 1, KZR-616 QW, 45 mg + SOC (Phase 1b) | Cohort 2, KZR-616 QW, 60 mg + SOC (Phase 1b) | Cohort 2a, KZR-616 QW, 30 mg x 2 Wks, 45 mg x 2 Wks, 60 mg x 9 Wks + SOC (Phase 1b) | Cohort 2b, KZR-616 QW, 30 mg x 1 wk, 60 mg x 12 Wks + SOC (Phase 1b) | Cohort 2c, KZR-616 QW, 30 mg x 1 wk, 60 mg x 12 Wks + SOC (Phase 1b) | Cohort 3, KZR-616 QW, 30 mg x 1 wk, 75 mg x 12 Wks + SOC (Phase 1b) | KZR-616 QW, 60 mg + SOC (Phase 2)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/5 | 0/14 | 0/6 | 0/8 | 0/6 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/5 | 2/14 | 1/6 | 0/8 | 0/6 | 2/22
Other Adverse Events (participants affected / at risk) | 8/8 | 5/5 | 12/14 | 4/6 | 7/8 | 3/6 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1, KZR-616 QW, 45 mg + SOC (Phase 1b) (N=8) | Cohort 2, KZR-616 QW, 60 mg + SOC (Phase 1b) (N=5) | Cohort 2a, KZR-616 QW, 30 mg x 2 Wks, 45 mg x 2 Wks, 60 mg x 9 Wks + SOC (Phase 1b) (N=14) | Cohort 2b, KZR-616 QW, 30 mg x 1 wk, 60 mg x 12 Wks + SOC (Phase 1b) (N=6) | Cohort 2c, KZR-616 QW, 30 mg x 1 wk, 60 mg x 12 Wks + SOC (Phase 1b) (N=8) | Cohort 3, KZR-616 QW, 30 mg x 1 wk, 75 mg x 12 Wks + SOC (Phase 1b) (N=6) | KZR-616 QW, 60 mg + SOC (Phase 2) (N=22)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1, KZR-616 QW, 45 mg + SOC (Phase 1b) (N=8) | Cohort 2, KZR-616 QW, 60 mg + SOC (Phase 1b) (N=5) | Cohort 2a, KZR-616 QW, 30 mg x 2 Wks, 45 mg x 2 Wks, 60 mg x 9 Wks + SOC (Phase 1b) (N=14) | Cohort 2b, KZR-616 QW, 30 mg x 1 wk, 60 mg x 12 Wks + SOC (Phase 1b) (N=6) | Cohort 2c, KZR-616 QW, 30 mg x 1 wk, 60 mg x 12 Wks + SOC (Phase 1b) (N=8) | Cohort 3, KZR-616 QW, 30 mg x 1 wk, 75 mg x 12 Wks + SOC (Phase 1b) (N=6) | KZR-616 QW, 60 mg + SOC (Phase 2) (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cataract nuclear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acid peptic disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (7) | 1 (1) | 5 (7)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (6) | 5 (8) | 1 (6) | 4 (24) | 3 (10) | 9 (22)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (7) | 3 (6) | 1 (3) | 2 (2) | 1 (1) | 9 (14)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (10)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (4) | 4 (9)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (13) | 0 (0) | 3 (19)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (16)
Injection site discolouration (General disorders) | 0 (0) | 1 (10) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Injection site erythema (General disorders) | 5 (30) | 2 (7) | 5 (16) | 2 (2) | 6 (58) | 0 (0) | 12 (66)
Injection site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site indentation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (12) | 5 (28)
Injection site mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (40)
Injection site nodule (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 4 (11) | 0 (0) | 0 (0) | 0 (0) | 6 (30)
Injection site pruritus (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (6)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 2 (7) | 0 (0) | 2 (3) | 0 (0) | 4 (31)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 3 (3)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 3 (10) | 1 (6) | 2 (5) | 3 (5) | 13 (45)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Selective IgG subclass deficiency (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis Escherichia coli (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post vaccination syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (16)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (41)
Differential white blood cell count abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram PR prolongation (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reticulocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (9)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (9) | 1 (2) | 1 (10) | 0 (0) | 5 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (12) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 1 (1) | 2 (13) | 3 (9) | 3 (11) | 2 (6) | 1 (3) | 11 (32)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Migraine with aura (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Pelvic cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (9) | 0 (0) | 3 (9)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
In Phase 2, of note, prior to the adoption of the open-label study design to improve enrollment after the onset of the COVID-19 pandemic, 1 patient with active proliferative LN was enrolled in Phase 2 under the earlier randomized, placebo-controlled, double-blind design. This patient was randomized to zetomipzomib at a dose of 30 mg SC weekly for 13 weeks and completed 12 of 13 dose administrations and all protocol-required procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall have the right to publish or present their own data resulting from the Study ("Publication") upon the earlier of: (a) the date following a multicenter publication coordinated by Sponsor regarding the Protocol; (b) 12 months after completion of the Protocol by all sites; or (c) the date after submission of the Study Data by Sponsor to the FDA.

The PI must furnish Sponsor with a copy of any Publication at least 30 days in advance of the proposed submission or presentation date.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT03393013/Prot_SAP_000.pdf